CLINICAL TRIAL: NCT03356444
Title: The Evaluation of First-line Treatment Efficacy of Docetaxel and Abiraterone in Metastatic Castration-resistant Prostate Cancer Patients With Intraductal Carcinoma of the Prostate and the Exploration of the Genes Related to Treatment Effect
Brief Title: Docetaxel Versus Abiraterone as First-line Treatment in mCRPC Patients With Intraductal Carcinoma of the Prostate
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Hao Zeng, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-16
Record Dates: First submitted 2017-11-09; First posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer; Castration-resistant Prostate Cancer; Drug
Keywords: abiraterone; docetaxel; Castration-resistant Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Docetaxel

STUDY DESIGN:
Masking Description: The administration methods of the two groups are different, therefore, the investigators decide not to use masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Abiraterone group (Experimental): Abiraterone acetate is administered in this arm.
  Interventions: Drug: Abiraterone Acetate
- Docetaxel group (Active Comparator): Docetaxel is administered in this arm.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone Acetate: orally, 1000mg, qd, plus with prednisone orally, 5mg, bid. Course of treatment: Stop the treatment until biochemical, clinical or radiographic progression occurs.
  Arms: Abiraterone group
Drug: Docetaxel — Docetaxel: intravenously, 75 mg/m^2, over 1 h every 3 weeks, plus with prednisone, orally, 10 mg, qd.
  Course of treatment: Stop the treatment until biochemical, clinical or radiographic progression occurs. If no progression, stop until 10 cycles of traetment
  Arms: Docetaxel group

SUMMARY:
Metastatic castration-resistant Prostate cancer (mCRPC) is a very late stage of prostate cancer with poor prognosis. Although there are several treatment strategies available for mCRPC, these drugs are not always effective for every patient. Also, it's still not clear what's the best therapeutic choice for a certain group of patients.

In the previous works of the investigators, a subtype of prostate cancer, intraductal carcinoma of the prostate (IDC-P) was studied. The investigators have reported in their two published papers that, IDC-P is an adverse pathological type associated with rapid disease progression. They also found in another study that, for patients with IDC-P, Abiraterone seemed to have better treatment efficacy than Docetaxel-based chemotherapy as first-line treatment for mCRPC, in terms of either PSA-response and PSA-progression free survival. So, in this study, the investigators hope to design a prospective study to verify the predictive ability of IDC-P in the first-line treatment of mCRPC.

With disease progression, the drug resistance will inevitably occur in all patients after the treatment of CRPC. However, the exact mechanism of this process is not yet known. So, in this study the investigators are also trying to explore some of the genes related to the treatment efficacy by means of the next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥40 years old
2. Positive IDC-P status confirmed by pathological examination.
3. Bone or visceral metastatic disease confirmed by image examination.
4. Castration resistant confirmed according to the criteria of 2014 EAU guidelines.
5. The ECOG score of the patient is ≤1
6. Expected survival over 3 months
7. Blood routine test: neutrophil ≥1.5 × 10^9, platelets >100 × 10^9 and hemoglobin ≥90g/L
8. Blood biochemical indexes: bilirubin≤1.5×Upper limit of normal; AST≤2.5×Upper limit of normal; serum creatinine≤1.5×Upper limit of normal; serum calcium≤12.0mg/dL.
9. Coagulation function: Prothrombin time ≤1.5×Upper limit of normal
10. The following diseases were not found within 12 months: myocardial infarction, severe or unstable angina pectoris, asymptomatic heart failure, cardiovascular and cerebrovascular accident or transient ischemic attack, etc.
11. All patients should sign informed consent.

Exclusion Criteria:

1. Patients who had other types of cancer besides prostate cancer were excluded.
2. Patients With non-acinar adenocarcinoma except intraductal carcinoma of the prostate, including ductal adenocarcinoma, neuroendocrine carcinoma or small cell carcinoma of the prostate.
3. Prior chemotherapy or abiraterone for the treatment of mCRPC.
4. Patients with renal decompensation requiring hemodialysis or peritoneal dialysis.
5. Patients with severe active clinical infection
6. Patients with coagulopathy or bleeding
7. Patients who received major surgery or severe trauma within the first 4 weeks before admission.
8. Patients with a history of allogeneic organ transplantation or bone marrow transplantation
9. Patients with known or suspected allergy to research drugs.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patient can enter this study
Enrollment: 140 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PSA-Progression free survival (PSA-PFS) | Up to 40 months
  PSA progression was defined as an increase in the PSA level of 25% or more above the nadir (and by ≥ 2 ng/ml), with confirmation of 4 or more weeks later.
Radiographic progression free survival (rPFS) | Up to 40 months
  rPFS was defined 1) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria; or 2) as at least two new lesions on first post-treatment bone scan, with at least two additional lesions on the next bone scan.

SECONDARY OUTCOMES:
PSA response rate | Up to 40 months
  PSA response is defined as ≥ 50% decline in PSA level from baseline, maintained for≥ 4 weeks
Overall survival (OS) | Up to 40 months
  OS was defined as the duration from the initiation of treatment to death of any cause
Eastern Cooperative Oncology Group (ECOG) score | Up to 40 months
  0 - Fully active, able to carry on all pre-disease performance without restriction;
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light house work, office work;
  2. - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours;
  3. - Capable of only limited self-care, confined to bed or chair more than 50% of waking hours;
  4. - Completely disabled. Cannot carry out on any self-care; totally confined to bed or chair.

IPD SHARING:
Plan to Share IPD: No